CLINICAL TRIAL: NCT07232823
Title: Brief Culturally Adapted Cognitive Behaviour Therapy (CaCBT) for Obsessive-Compulsive Disorder: A Randomised Controlled Trial From Pakistan
Brief Title: Brief Culturally Adapted CBT for OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CaCBTOCD24
Record Dates: First submitted 2024-10-16; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Obsessive-Compulsive Disorder; Cognitive Behavioral Therapy
Keywords: CBT; CaCBT; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: This will be a randomised, controlled, assessor-blind clinical trial. It will be carried out at Recovery Psychiatric & Addiction Treatment, Rehab & Psychotherapy Centre, Lahore, and Dr Muhammad Afzal Khan Clinic, Faisalabad. The participants will be provided with oral and written information about the study, and written informed consent will be obtained. Participants who agree to participate will be allocated to one of the groups: brief CaCBT plus TAU (Treatment group) or TAU alone (Control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief culturally adapted CBT (CaCBT) group (Experimental): Participants in this group will receive the Culturally Adapted CBT (CaCBT) manual along with treatment as usual (which typically involves medication prescriptions and regular hospital visits). The manual will focus on psychoeducation, symptom management, Exposure and Response prevention (ERP), thought distraction techniques, relaxation exercises, detection of mood and thoughts, cognitive errors, changing negative thinking, behavioural activation, problem solving, improving relationships and communication skills, Thought diaries and progress diary.
  Interventions: Other: Brief culturally adapted cognitive behaviour therapy (CaCBT)
- Treatment as usual group (No Intervention): Participants in this group will receive only treatment as usual (TAU), which typically involves medication prescriptions and regular hospital visits. Research psychologists delivering the intervention will not be involved with participants allocated to TAU.

INTERVENTIONS:
Other: Brief culturally adapted cognitive behaviour therapy (CaCBT) — The intervention will focus on psychoeducation, symptom management, Exposure and Response prevention (ERP), thought distraction techniques, relaxation exercises, detection of mood and thoughts, cognitive errors, changing negative thinking, behavioural activation, problem solving, improving relationships and communication skills, Thought diaries and progress diary.
  Arms: Brief culturally adapted CBT (CaCBT) group

SUMMARY:
The purpose aims to assess the efficacy of Brief Culturally Adapted Cognitive Behaviour Therapy (Ca-CBT) for the treatment of Obsessive Compulsive Disorder (OCD).

DETAILED DESCRIPTION:
The presence of obsessions and compulsions characterises obsessive-compulsive disorder (OCD). Obsessions are intrusive, unwanted thoughts, images, or impulses that are distressing and difficult to control. These obsessive thoughts cause significant emotional discomfort. Conversely, compulsions are repetitive behaviours or mental acts performed in response to an obsession or according to rigid rules. These actions are intended to reduce anxiety or prevent a feared event, even though they may not logically connect to the feared outcome. The individual often experiences temporary relief from distress through these ritualistic responses despite their lack of practical relevance to the obsessive fears.

Cognitive Behaviour Therapy (CBT) is widely recognised as a treatment option in both the US and UK National Treatment Guidelines (National Institute for Health and Care Excellence, 2009; American Psychiatric Association, 1993). There is strong evidence supporting CBT's effectiveness in treating, preventing relapse, and managing depression and anxiety (Embling, 2002; Fava et al., 1998; Paykel et al., 1999; Thase, 1997).

However, despite this evidence, there has been limited progress in assessing CBT's effectiveness in low and middle-income countries. CBT may require adaptation in non-Western cultures, as it involves exploring and modifying automatic thoughts and core beliefs (Padesky and Greenberger, 1995).

Preliminary research suggests that treatment manuals based on fundamental CBT principles are effective (Husain et al., 2013; Rahman et al., 2008; Sumathipala et al., 2008; Araya et al., 2003). In Pakistan, an adapted version of CBT for depression was conducted, demonstrating its effectiveness in primary care settings (Naeem et al., 2011). Similarly, a pilot study was conducted on brief culturally adapted cognitive behaviour therapy for obsessive-compulsive disorder (Aslam et al. 2015).

This study aims to conduct a randomised controlled trial using brief culturally adapted cognitive behaviour therapy for obsessive-compulsive disorder in Pakistan, as limited research is available on this aspect. Conducting this trial can provide valuable data on the effectiveness of culturally adapted CBT in the Pakistani cultural setting, informing both local and international practices.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or above
* Participants with at least an elementary level of reading and writing
* Clinical diagnosis of Obsessive Compulsive Disorder, either alone or comorbid with depression or anxiety

Exclusion Criteria:

* Participants with excessive use of alcohol or drugs (using ICD-10 RDC for alcohol or drug abuse or dependence)
* Those with significant cognitive impairment (for example, intellectual disability or dementia)
* Or those with OCD comorbid active psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of brief culturally adapted cognitive behaviour therapy (CaCBT) for OCD | 6 weeks
  By comparing pre- and post-treatment OCD scores measured through the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS).
Acceptability of the brief culturally adapted cognitive behaviour therapy (CaCBT) for OCD | 6 weeks
  Feedback will be taken from both patients and their family members, who will be trained as co-therapists, to evaluate their satisfaction with the therapy.

SECONDARY OUTCOMES:
Reduction in depression and anxiety associated with OCD | 6 weeks
  By comparing pre- and post-treatment depression and anxiety scores measured through the Hospital Anxiety and Depression Scale (HADS).
Reduction in functioning decline associated with OCD | 6 weeks
  By comparing pre- and post-treatment scores on the Brief Disability Questionnaire (BDQ).

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, Principal Investigator — Professional Association of Cognitive Therapy; Muhammad Aslam, Principal Investigator — Professional Association of Cognitive Therapy
Locations (1):
- Professional Association of Cognitive Therapy, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided